CLINICAL TRIAL: NCT06201520
Title: The Effect of Acupuncture and Laser Acupuncture for Carpal Tunnel Syndrome-A 3-arm, Randomized Sham Laser Acupuncture Controlled Study
Brief Title: The Effect of Acupuncture and Laser Acupuncture for Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901768A3
Record Dates: First submitted 2021-08-17; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome; Acupuncture; Laser Acupuncture
Keywords: Carpal Tunnel Syndrome; Acupuncture; Laser Acupuncture
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MA group (manual acupuncture group) (Experimental): Acupunctue Needle: 1 inch- 32 gauge（0.3x25 mm）for 20 min after De-qi Acupoints selection: PC4[Ximen], PC6[Neiguan], PC7[Daling], PC8[Laogong], HT2[Qingling], HT7[Shenmen], HT8[Shaofu], LU9[Taiyuan], LI11[Quchi]
  Interventions: Procedure: manual acupuncture; Device: wrist splint
- LA group (laser acupuncture group) (Experimental): laser acupuncture gruoup with LaserPen, 150 mW; wavelength, 810nm; area of probe, 0.03cm2; power density, 5W/cm2; pulsed wave; Nogier C frequency for 4 J each points The acupoints selection is the same as the MA group.
  Interventions: Device: laser acupuncture; Device: wrist splint
- SLA group (sham laser acupuncture group) (Sham Comparator): sham laser acupuncture group is designed with the same acupoints selection and no energy output
  Interventions: Device: sham laser acupuncture; Device: wrist splint

INTERVENTIONS:
Procedure: manual acupuncture — manual acupuncture
  Arms: MA group (manual acupuncture group)
Device: laser acupuncture — laser acupuncture therapy
  Arms: LA group (laser acupuncture group)
Device: sham laser acupuncture — sham laser acupuncture
  Arms: SLA group (sham laser acupuncture group)
Device: wrist splint — wear wrist splint at night

SUMMARY:
Acupuncture and laser acupuncture treatments have been proven to be effective and safe treatments for carpal tunnel syndrome(CTS). However, there is still a lack of direct comparative studies of acupuncture and laser acupuncture in the treatment of CTS. A 3-arm, randomized controlled study in acupuncture, laser acupuncture study and sham laser acupuncture therapy was designed for patient with carpal tunnel syndrome. The Glabal symptom score (GSS), Boston Carpal Tunnel Questionnaire (BCTQ), neurophysiological study, morphological examination under ultrasonography will be evaluated before and after treatment. Comparison of therapeutic efficacy of acupuncture, laser acupuncture and sham laser acupuncture in the treatment of CTS will be explored.

DETAILED DESCRIPTION:
The primary outcome will analyze the change of the Glabal symptom score (GSS) during intervention peroid. The secondary outcome will evaluate the neurophysiological study, morphological examination under ultrasonography before and after treatment. Comparison of therapeutic efficacy of acupuncture, laser acupuncture and sham laser acupuncture in the treatment of CTS will be explored.

ELIGIBILITY:
Inclusion Criteria:

* patients with mild to moderate carpal tunnel syndrome diagnosed by neurophysiological examination
* symptoms of carpal tunnel syndrome such as pain and numbness
* those who are willing to sign informed consent form for subjects

Exclusion Criteria:

* (1) Those who have not signed the informed consent
* (2) Patients diagnosed with severe carpal tunnel syndrome
* (3) Those who have had a history of surgery on their hands and palms
* (4) Space-occupying lesions such as tumors, bone spurs, synovial membrane tissue hypertrophy, etc.
* (5) People with a history of diabetes, rheumatoid arthritis, and hypothyroidism (HbA1c>6.5, RF positive, Free T4, TSH in abnormal range)
* (6) Patients with end-stage renal disease
* (7) Pregnant and alcoholic patients
* (8) Polyneuropathy patients
* (9) Clinical symptoms with C6~8 cervical radiculopathy
* (10) Those who are obviously infected
* (11) Those with a serious illness requiring hospitalization

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The Boston Carpal Tunnel Questionnaire(BCTQ) changes | from baseline to 3 months
  The Boston Carpal Tunnel Questionnaire(BCTQ) is a questionnaire for CTS patients, which has been used widely in the world. It contains two parts. One part is the symptom severity scale (BCTQsss) which contains eleven questions about symptom severity, and another part is the function severity scale (BCTQfss) contains eight questions about functional status evaluation. Each selection option includes 1~5 to present different degrees of severity ("5" is the most severe). The max of BCTQsss is 55 and the min is 11. The max of BCTQfss is 40 and the min is 8. The higher scores mean a worse outcome.
Global symptoms score(GSS) changes | from baseline to 3 months
  GSS is a questionnaire to evaluate the severity of five symptoms, including pain, numbness, paresthesias, weakness/ clumsy, and nocturnal awakening for CTS patients.
  The score of pain, numbness, and paresthesias according to the magnitude: from 0 (nil) to 10 (most severe).
  The score for weakness/ clumsiness is according to the severity: 0 (none); 2(mild); 3(moderate); 4(severe); 5(very severe).
  The score for nocturnal awakening is according to how many times awaked in one week: 0(never); 2(once or twice); 4(three or four times); 6(five to seven times); 8(eight to ten times); 10(more than ten times).
  The total score added up forms the GSS score. The minimum score is 0, and the maximum score is 50. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
compound motor action potential(CMAP) | from baseline to 3 months
  Nerve Electrophysiological examination of median nerve.The neurophysiological study of the median nerve will be recorded and compared before and after 15 sessions of treatments including compound motor action potential(CMAP).
  The unit of CMAP is millivolt (mV).
motor distal latency(MDL) | from baseline to 3 months
  Nerve Electrophysiological examination of median nerve. The neurophysiological study of the median nerve will be recorded and compared before and after 15 sessions of treatments including motor distal latency(MDL).
  The unit of motor distal latency is millisecond (ms).
Sensory nerve action potential (SNAP) | from baseline to 3 months
  Nerve Electrophysiological examination of median nerve. The neurophysiological study of the median nerve will be recorded and compared before and after 15 sessions of treatments including Sensory nerve action potential (SNAP).
  The unit of SNAP is also millivolt (mV).
sensory distal latency(SDL) | from baseline to 3 months
  Nerve Electrophysiological examination of median nerve. The neurophysiological study of the median nerve will be recorded and compared before and after 15 sessions of treatments including sensory distal latency(SDL).
  The unit of sensory distal latency is also millisecond (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Huang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maeda Y, Kim H, Kettner N, Kim J, Cina S, Malatesta C, Gerber J, McManus C, Ong-Sutherland R, Mezzacappa P, Libby A, Mawla I, Morse LR, Kaptchuk TJ, Audette J, Napadow V. Rewiring the primary somatosensory cortex in carpal tunnel syndrome with acupuncture. Brain. 2017 Apr 1;140(4):914-927. doi: 10.1093/brain/awx015. PMID 28334999
- [Result] Hadianfard M, Bazrafshan E, Momeninejad H, Jahani N. Efficacies of Acupuncture and Anti-inflammatory Treatment for Carpal Tunnel Syndrome. J Acupunct Meridian Stud. 2015 Oct;8(5):229-35. doi: 10.1016/j.jams.2014.11.005. Epub 2014 Nov 29. PMID 26433799
- [Result] Chen CC, Wu YT, Su YC, Shen YP, Chen FP. Efficacy of laser acupuncture for carpal tunnel syndrome: A study protocol for a prospective double-blind randomized controlled trial. Medicine (Baltimore). 2019 Jul;98(30):e16516. doi: 10.1097/MD.0000000000016516. PMID 31348263